CLINICAL TRIAL: NCT04043546
Title: Observational Feasability Study of Home-based Training With Therabands in PAD-patients - Addressing the Uncertainty of Acceptance, Satisfaction and Usability of a Home-based, Tele-monitored Program Combining Aerobic and Resistance Components in PAD-patients.
Brief Title: Observational Feasibility Study of Home-based Training With Therabands in PAD-patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Roselien Buys, Principal Investigator, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAD-feasibility
Record Dates: First submitted 2018-07-10; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Peripheral Artery Disease; Intermittent Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Intervention Model Description: Patients enrolled in the study receive a novel physiotherapy program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise intervention (Experimental)
  Interventions: Behavioral: aerobic+resistance exercise training program

INTERVENTIONS:
Behavioral: aerobic+resistance exercise training program — Personalized exercise program based on the inclusion testing and patient screening will be provided to the patient. The program will consist of a gradual walking program as well as a gradual resistance training program using therabands.

SUMMARY:
The study is an observational feasibility study to evaluate the feasibility of a combined aerobic+resistance training program in patients with IC.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 50 yrs;
* ankle-brachial index (ABI) ≤ 0.9 in one or two legs;
* Fontaine stage II (Rutherford I 1-3) of PAD (new onset or conservatively treated);
* body mass index <35 kg/m 2 ;
* resting systolic blood pressure (BP) <160 mmHg and diastolic BP <105 mmHg;
* ability to walk at least 2 min at 2.0 mph;
* ability to undertake an incremental treadmill test;
* decrease of at least 15% in ABI after a maximal treadmill test;
* not currently engaging in any regular exercise program.

Exclusion Criteria:

* exercise induced signs of myocardial ischemia or complex ventricular arrhythmias;
* no access to laptop or internet;
* no medical clearance for exercise

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
user satisfaction | 4 weeks
  self-developed questionnaire based evaluation of user satisfaction
walking distance | 4 weeks
  pain free and maximal walking distance are recorded using the Gardner treadmill protocol.

SECONDARY OUTCOMES:
Physical activity | 2 months
  Physical activity, defined total active energy expenditure (kcal) is obtained from objective measurement of physical activity during 7 consecutive days using the Sensewear device.

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cornelis N, Buys R, Dewit T, Benoit D, Claes J, Fourneau I, Cornelissen V. Satisfaction and Acceptability of Telemonitored Home-Based Exercise in Patients With Intermittent Claudication: Pragmatic Observational Pilot Study. JMIR Rehabil Assist Technol. 2021 Mar 22;8(1):e18739. doi: 10.2196/18739. PMID 33749616